CLINICAL TRIAL: NCT02691442
Title: Comparison of the Analgesic Effect of the Local Anesthetics Ropicacaine, Levobupivacaine, and Levobupivacaine + Epinephrin Via Interscalene Nerve Block in Patients Undergoing Shoulder Arthroscopy Under General Anesthesia
Brief Title: Comparison of the Analgesic Effect of Different Local Anesthetics in Interscalene Nerve Block for Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, MD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC 10/45/315
Record Dates: First submitted 2016-02-01; First posted 2016-02-25 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Other Peripheral Nerve Disease
Keywords: Peripheral nerve block
MeSH Terms: interventions — Ropivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine 0.75% (Active Comparator): The investigators administer 5 milliliters of Ropivacaine 0.75% in the inter scalene space
  Interventions: Drug: Ropivacaine 0.75%
- Levobupivacaine 0.5% (Active Comparator): The investigators administer 5ml of Levobupivacaine 0.5% in the inter scalene space
  Interventions: Drug: Levobupivacaine 0.5%
- Levobupivacaine 0.5% + epinephrin (Active Comparator): The investigators administer 5ml of Levobupivacaine 0.5% + epinephrin 1/200000 in the inter scalene space
  Interventions: Drug: Levobupivacaine 0.5% + epinephrin 1/200000

INTERVENTIONS:
Drug: Ropivacaine 0.75% — The investigators adminster 5ml of Ropivacaine 0.75% in an ultrasound-guided inter scalene nerve block
  Other Names: Naropin
  Arms: Ropivacaine 0.75%
Drug: Levobupivacaine 0.5% — The investigators adminster 5ml of Levobupivacaine 0.5% in an ultrasound-guided inter scalene nerve block
  Other Names: Chirocaine
  Arms: Levobupivacaine 0.5%
Drug: Levobupivacaine 0.5% + epinephrin 1/200000 — The investigators adminster 5ml of Levobupivacaine 0.5% + epinephrin 1/200000 in an ultrasound-guided inter scalene nerve block
  Other Names: Chirocaine
  Arms: Levobupivacaine 0.5% + epinephrin

SUMMARY:
Several reports have compared the duration of action of levobupivacaine and ropivacaine as local anesthetic. The most widely used method for sensory function evaluation is though means of a pinprick test. The investigators want to use the novel method of Quantitative Sensory Testing to better evaluate the anesthetic activity. This method used hot and cold sensation to assess small nerve fiber function. The investigators will assess the duration of action of different drugs when used in an inter scalene nerve block in patients scheduled for shoulder surgery.

DETAILED DESCRIPTION:
This study aims to compare the length of the analgesic effect of different local anesthesic solutions, used in an interscalene nerve block. This will be objectified by measuring the changes in small nerve functioning, using quantative sensory testing. Based on the results of a previous study, the investigators reduce the dose of the administered local anesthetic, expecting a similar length of action using these smaller doses.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia class I or II
* Scheduled for shoulder surgery

Exclusion Criteria:

* Mental retardation
* Allergy for local anesthetics
* NSAID intolerance or contraindicated
* Diabetes mellitus
* Chronic use of pain killers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Length of nerve block measured in longitudinally recorded significant changes in sensory thresholds using quantitative sensory testing | 24 hours after intervention
  Length of difference in cold and heat pain and sensation measured with quantitative sensory testing

SECONDARY OUTCOMES:
Need for rescue drugs, as requested by the patient after surgery | 24 hours after intervention
Motor activity block, longitudinally recorded inability to move the blocked limb | 24 hours after intervention
Intensity of nerve block, recorded as maximal changes in sensory thresholds using quantitative sensory testing | 24 hours after intervention
  The difference in threshold of cold and heat pain and sensation measured with quantitative sensory testing

CONTACTS AND LOCATIONS:
Overall Officials: Luc Serieus, MD, Study Chair — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sermeus LA, Schepens T, Hans GH, Morrison SG, Wouters K, Breebaart MB, Smitz CJ, Vercauteren MP. A low dose of three local anesthetic solutions for interscalene blockade tested by thermal quantitative sensory testing: a randomized controlled trial. J Clin Monit Comput. 2019 Apr;33(2):307-316. doi: 10.1007/s10877-018-0150-3. Epub 2018 May 3. PMID 29725795